CLINICAL TRIAL: NCT04670328
Title: Role of Hematological Parameters in the Stratification of COVID-19 Disease Severity
Status: Completed | Type: Observational
Sponsor: FMH College of Medicine and Dentistry (Other)
Responsible Party: Principal Investigator, Sadia Taj, Assistant Professor, FMH College of Medicine and Dentistry
Other Study IDs: FMHCMD
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Covid-19 disease; Neutrophil to Lymphocyte ratio; hematological manifestations
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — blood test
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Covid-19 disease severity: Mild, moderate, severe and critical disease
  Interventions: Diagnostic Test: not required

INTERVENTIONS:
Diagnostic Test: not required — Diagnostic tests( hematological parameters) were assessed.

SUMMARY:
The hemostatic abnormalities in COVID-19 are related with disease progression, severity and mortality. The Objective of our study is to evaluate the role of hematological parameters in determination of COVID-19 disease severity.

DETAILED DESCRIPTION:
Objective:

COVID-19 virus involves respiratory as well as other body systems including cardiovascular, gastrointestinal, neurological, immunological and hematopoietic system. Patient of covid-19 pneumonia presents with wide range of hemostatic abnormalities. These hemostatic abnormalities in COVID-19 are related with disease progression, severity and mortality. The Objective of our study is to evaluate the role of hematological parameters in determination of COVID-19 disease severity.

Material and Method:

This was a retrospective study, conducted in Department of Pathology and Department of medicine, FMH college of Medicine and Dentistry from May 2020 to July 2020. Total of 101, confirmed cases of covid-19 disease, both genders between 17 to 75-year age were included. Hematological parameters were compared in mild, moderate, severe and critical disease group. Continuous variables were analyzed by using non parametric, Kruskal Wallis test while categorical variables were analyzed by chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed cases of covid-19 disease
* Both genders
* 17 to 75 year age

Exclusion Criteria:

* known case of chronic liver disease
* known hematological diseases were excluded

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: diagnosed cases of covid-19
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
complete blood count- Hemoglobin. White blood count, platelet count, Neutrophil to lymphocyte ratio | 3 months
  disease severity was assessed on basis of hematological parameters.

SECONDARY OUTCOMES:
PT, APTT and D-dimer | 3 months
  improvement in PT, APTT and D-dimer levels were assessed

OTHER OUTCOMES:
LDH, serum ferritin level | 3 months
  improvement in LDH and were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Ayaz Lone, MBBS,FCPS, Study Chair — FMH College of Medicine and Dentistry
Locations (1):
- FMH college of medicine and dentistry, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD